CLINICAL TRIAL: NCT04926467
Title: An Open Label, Phase II Study of Chemotherapy + Anakinra in Patients With Resectable, Locally Advanced or Potentially Resectable Pancreatic Adenocarcinoma (PDAC)
Brief Title: Chemotherapy + Anakinra in Patients With Pancreatic Adenocarcinoma (PDAC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020-476
Record Dates: First submitted 2021-06-01; First posted 2021-06-15 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Adenocarcinoma
MeSH Terms: interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Anakinra plus Chemotherapy (Experimental): Patients will receive Anakinra during both pre-operative chemotherapy with Nab-paclitaxel, gemcitabine and cisplatin, followed by surgery and post-operative chemotherapy with 5-fluorouracil, oxaliplatin, and irinotecan.
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — Anakinra (100 mg) twice a day (BID), daily, will be self-administered subcutaneously starting on D1 of chemotherapy. Anakinra will be held 2 days prior to surgery. A dosing diary will be given to the patient for anakinra documentation.
  Other Names: Kineret

SUMMARY:
Based on a central role of inflammation in pancreas cancer, the role of IL 1 in acute and chronic inflammation , the inhibitory effect of IL 1 alfa and beta by anakinra and preliminary experience with anakinra in combination with chemotherapy in metastasis (with FOLFIRINOX) and localized disease (with gemcitabine/abraxane/cisplatin), a phase 2 study with anakinra in combination with perioperative chemotherapy for patients with PDAC is being proposed.

DETAILED DESCRIPTION:
This is an open-label, single-arm, prospective phase II study conducted by Baylor Scott and White Research Institute in Dallas.

The study will enroll patients with pancreatic adenocarcinoma that are planned to receive pre-operative chemotherapy followed by surgical resection and post operative treatment. Local surgical/biopsy and pathology reports will constitute adequate documentation of histology/cytology for study inclusion.

Patients will receive pre- and post-operative chemotherapy plus Anakinra. Specifically, the pre-operative chemotherapy regimen will be a combination of Nab-paclitaxel, gemcitabine and cisplatin, while post-operative chemotherapy will use 5-Fluorouracil, oxaliplatin, and irinotecan. Patients will also receive growth factor (Neupogen followed by Neulasta) for safety and to ensure that treatment is not delayed due to neutropenic effects of chemotherapy.

Anakinra will be self-administered by the participants through out the treatment period. A treatment break of 2 days will be given prior to the surgery day.

ELIGIBILITY:
Inclusion Criteria:

* A patient will be eligible for inclusion in this study if he or she meets all of the following criteria:

  1. 18 years of age or older
  2. Histologically or Cytologically confirmed pancreatic ductal adenocarcinoma. Mixed subtypes of adenocarcinoma are acceptable as long as majority of cells are ductal adenocarcinoma.
  3. Resectable, locally advanced or potentially resectable pancreatic adenocarcinoma
  4. American Joint Committee on Cancer (AJCC) Stage I-III Pancreatic carcinoma.
  5. Patient has Eastern Cooperative Oncology Group( ECOG ) Performance Status 0 to 1
  6. Serum albumin ≥2.0 g/dL.
  7. Adequate hematologic function as defined by:

     1. Absolute neutrophil count (ANC) ≥1500/mm3;
     2. Platelets ≥70,000 x 10^3/µl;
     3. Hemoglobin ≥9 g/dL (in the absence of red blood transfusion).
  8. Adequate liver function, as defined by:

     1. Serum total bilirubin ≤2 x ULN mg/dL, prior to initiation of treatment.
     2. ALT (SGPT) and AST (SGOT) ≤2.5 x upper limit of normal (ULN).
  9. Adequate renal function, as defined by serum creatinine≤ 1.5 x ULN, or creatinine clearance ≥50 mL/min
  10. Women of child bearing potential and men must agree to use contraception throughout the study and for one month after the last anakinra administration.
  11. Subjects must understand and sign the informed consent form
  12. Patients must be accessible for treatment and follow-up.

Exclusion Criteria:

* A patient will be ineligible for inclusion in this study if he or she meets any of the following criteria:

  1. <18 years of age
  2. History of organ transplant.
  3. Patients with islet cell neoplasms
  4. Patients with stage IV pancreatic carcinoma
  5. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
  6. Known active infection with hepatitis B or hepatitis C
  7. Presence of clinically significant cirrhosis as determined by the investigator
  8. Known HIV positive status.
  9. Current, active immunosuppressive therapy such as cyclosporine, tacrolimus, etc.
  10. Major surgery or vascular device placement within 2 weeks prior to Day 1 of treatment in study
  11. Prior chemotherapy or radiation for pancreatic cancer
  12. History of allergy or hypersensitivity to the study drugs
  13. Patient is enrolled in any outside therapeutic clinical protocol or investigational trial with an investigational drug within 5 half-lives prior to Study ID assignment
  14. Previous or current treatment with anakinra, canakinumab or any other IL-1 inhibitor
  15. Other malignancy within five years(except cutaneous, non-melanoma malignancies or cervical carcinoma in site), unless the probability of recurrence of the prior malignancy is <5% as determined by the Principal Investigator based on available information.
  16. Significant cardiac disease (uncontrolled congestive heart failure (CHF), myocardial infarction or significant ventricular arrhythmias) within the last six months.
  17. Other severe and/or uncontrolled medical conditions (e.g: prior gastrointestinal (GI) disease or history of prior pelvic or abdominal radiation) or other conditions deemed by investigator as unsuitable for participation/enrollment
  18. Peripheral sensory neuropathy > or equal to grade 2 at baseline
  19. Abnormal liver function tests as follows:

      1. Total bilirubin of > 2 x ULN
      2. AST or ALT > 5x ULN
  20. Serum albumin ˂ 2.0 g/dL.
  21. Abnormal hematologic function as follows :

      1. Absolute neutrophil count (ANC) ˂ 1500/mm3;
      2. Platelets ˂ 70,000 x 10^3/µl;
      3. Hemoglobin ˂ 9 g/dL (in the absence of red blood transfusion).
  22. Pregnant or nursing women
  23. No signed Informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-07-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
To determine the percentage of patients that have a normalization of CA19-9 after pre-op treatment with the combination of nab-paclitaxel (abraxane), gemcitabine, cisplatin and anakinra. | 24 months

SECONDARY OUTCOMES:
To determine the effect of anakinra in combination with perioperative chemotherapy on overall survival (OS) of PDAC patients. A benchmark of 24 months OS will be used to determine how many patients meet or exceed this goal. | 24 months
To determine the effect of anakinra in combination with perioperative chemotherapy on the median disease free survival (DFS). A benchmark of 12 months DFS will be used to determine how many patients meet or exceed this goal. | 12 months
To determine the effect of anakinra in combination with perioperative chemotherapy on response rate | 24 months
To determine the R0 resection rates (complete tumor removal with negative resection margins) obtained with anakinra + pre-operative chemotherapy. | 24 months
To describe the effect of anakinra in combination with perioperative chemotherapy on the prevalence and severity of pain by monitoring patients' pain level using memorial pain assessment card (MPAC). | 24 months
To determine the effect of anakinra in combination with perioperative chemotherapy on patients' health-related quality of life by monitoring patients using EORTC quality of life survey questionnaire (EORTC QLQ-C30). | 24 months
To determine the effect of anakinra in combination with perioperative chemotherapy on the inflammasomes ( IL6, CRP, IL1α and IL1β) in blood and in the resected pathology specimens. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: A. Scott Paulson, MD, Principal Investigator — Charles A. Sammons Cancer Center/Texas Oncology
Locations (1):
- Baylor University Medical Center, Charles A Sammons Cancer Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No